CLINICAL TRIAL: NCT05948137
Title: A Prospective Comparative Study of 18F-FDOPA PET/CT Versus 123I-MIBG Scintigraphy With SPECT/CT for the Diagnosis of Pheochromocytoma and Paraganglioma
Brief Title: F-18 FDOPA PET/CT Versus I-123 MIBG Scintigraphy With SPECT/CT for the Diagnosis of Pheochromocytoma and Paraganglioma
Status: Terminated | Type: Observational
Why Stopped: The study had to be prematurely stopped, falling short of the initial target due to prolonged shortages in the supply of 123I-MIBG.
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Sook Ryu, Professor, Asan Medical Center
Other Study IDs: FDOPA_2014_0901
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Pheochromocytoma; Paraganglioma
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pheochromocytoma / paraganglioma
  Interventions: Diagnostic Test: F-18 FDOPA PET/CT

INTERVENTIONS:
Diagnostic Test: F-18 FDOPA PET/CT — Nuclear medicine imaging modalities
  Other Names: I-123 MIBG SPECT/CT

SUMMARY:
Pheochromocytomas and paragangliomas (PPGLs) are chromaffin cells-derived tomours that originate from the adrenal medulla (80~85%) and the extra-adrenal sympathetic paraganglia in thorax, abdomen and pelvis (15~20%) or parasympathetic paraganglia in the head and neck region (~1%), respectively. Functional imaging, such as 123I-Meta-Iodobenzylguanidine (MIBG) scintigraphy with single photon emission computed tomography with a CT (SPECT/CT), offers high specificity for PPGL but necessitates 24-hour delayed imaging, pre-processing thyroid protection with a potassium iodide solution, and medication reconciliation to prevent the inhibition of 123I-MIBG uptake. Conversely, 18F-L-dihydroxyphenylalanine (FDOPA), a radiopharmaceutical for positron emission tomography (PET) imaging, is specifically absorbed and accumulated by chromaffin cells, offering better image quality and convenience compared to 123I-MIBG scintigraphy. 18F-FDOPA PET/CT has been approved for the localization, staging, and detection of PPGL recurrences in European and other countries. Therefore, the aim of this study was to compare prospectively the diagnostic performances of 18F-FDOPA PET/CT and 123I-MIBG scintigraphy with SPECT/CT in patients with PPGL.

ELIGIBILITY:
Inclusion Criteria:

1. suspected PPGL based on a biochemical screening, including 24-hour urinary total normetanephrine, metanephrine, norepinephrine, and epinephrine, along with plasma free concentrations of normetanephrine and metanephrine conducted within the past 6 months
2. an adrenal incidentaloma, suggestive of PPGL on anatomical imaging (CT or MRI) performed within the past 6 months
3. characteristic symptoms and signs of PPGL
4. suspected of recurrence or metastases of known PPGL.

Exclusion Criteria:

* pregnant and lactating women
* individuals aged less than 15 years
* patients with a serum creatinine level greater than 3 mg/dL due to chronic renal failure
* patients with a second primary cancer that was not in complete remission

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suspected of having PPGL or those showing recurrence and/or distant metastasis of PPGL were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Non-inferiority in diagnostic sensitivity of F-18 FDOPA PET/CT compared with that of I-123 MIBG SPECT/CT | Time interval of two imaging modalities was in the range of 1-15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No